CLINICAL TRIAL: NCT03199118
Title: The Use of Coronally Advanced Flap and Subepithelial Connective Tissue Graft With or Without Platelet Rich Fibrin in the Treatment of Miller Class I or II Gingival Recession: a Randomized Clinical Trial
Brief Title: Use of Platelet Rich Fibrin in Addition to CAF and SCTG for Treatment of Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Elbanna, Assistant lecturer in the oral medicine and periodontology department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sarahelbanna84
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Gingival Recession
Keywords: root coverage
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF+SCTG+PRF (Experimental): The patients suffering from class I or II gingival recession in the intervention group will receive a subepithelial connective tissue graft (SCTG) covered by platelet rich fibrin membrane (PRF) followed by a coronally advanced flap (CAF)
  Interventions: Procedure: CAF +SCTG; Other: platelet rich fibrin
- CAF+SCTG (Active Comparator): Control group patients with class I or II gingival recession will receive treatment that consists of CAF+SCTG only
  Interventions: Procedure: CAF +SCTG

INTERVENTIONS:
Procedure: CAF +SCTG — the use of coronally advanced flap (CAF) with sub-epithelial connective tissue graft (SCTG) from the palate to cover gingival recession
  Other Names: CTG
Other: platelet rich fibrin — in addition to coronally advanced flap and sub-epithelial connective tissue graft, PRF is also used in the surgical procedure to cover gingival recession
  Other Names: PRF
  Arms: CAF+SCTG+PRF

SUMMARY:
This research will be conducted in an attempt to achieve complete root coverage with physiologic probing depth and a harmonious view with the adjacent tissues using Platelet rich fibrin in conjunction with Coronally advanced flap and subepithelial connective tissue graft.

DETAILED DESCRIPTION:
The study population will be divided into 2 groups:

Group 1:

Patients suffering from Miller class I or II gingival recession will be treated with a coronally advanced flap in conjunction with a sub-epithelial connective tissue graft. The patients should be non-smoker, medically free and above 18 years

Group 2:

Patients suffering from Miller class I or II gingival recession will be treated with a coronally advanced flap in conjunction with a sub-epithelial connective tissue graft and platelet rich fibrin. the patients should meet the same inclusion criteria mentionned above.

ELIGIBILITY:
Inclusion Criteria:

- 1) Patients 18 years and older 2) Buccal recession defects classified as either Miller class I or II gingival recession.

3) Clinical indication and/or patient request for recession coverage 4) Good oral hygiene

Exclusion Criteria:

- 1) Miller Class III and IV gingival recession. 2) Any systemic diseases or any medication. 3) Pregnancy. 4) Patients undergoing radiotherapy. 5) Handicapped and mentally retarded patients. 6) Current and former smokers as smoking is a contra-indication for plastic periodontal surgery .

7) Teeth with cervical restorations, abrasion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azza Ezzelarab, Study Director — Professor of periodontics, Faculty of dentistry, Cairo university; Noha Ghallab, Study Director — Professor of periodontics, Faculty of dentistry, Cairo university
Locations (1):
- Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berlucchi I, Francetti L, Del Fabbro M, Testori T, Weinstein RL. Enamel matrix proteins (Emdogain) in combination with coronally advanced flap or subepithelial connective tissue graft in the treatment of shallow gingival recessions. Int J Periodontics Restorative Dent. 2002 Dec;22(6):583-93. PMID 12516830
- [Background] Bruno JF. Connective tissue graft technique assuring wide root coverage. Int J Periodontics Restorative Dent. 1994 Apr;14(2):126-37. PMID 7928129
- [Background] Gonshor A. Technique for producing platelet-rich plasma and platelet concentrate: background and process. Int J Periodontics Restorative Dent. 2002 Dec;22(6):547-57. PMID 12516826
- [Background] Keceli HG, Kamak G, Erdemir EO, Evginer MS, Dolgun A. The Adjunctive Effect of Platelet-Rich Fibrin to Connective Tissue Graft in the Treatment of Buccal Recession Defects: Results of a Randomized, Parallel-Group Controlled Trial. J Periodontol. 2015 Nov;86(11):1221-30. doi: 10.1902/jop.2015.150015. Epub 2015 Jul 16. PMID 26177630
- [Background] Marx RE, Carlson ER, Eichstaedt RM, Schimmele SR, Strauss JE, Georgeff KR. Platelet-rich plasma: Growth factor enhancement for bone grafts. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Jun;85(6):638-46. doi: 10.1016/s1079-2104(98)90029-4. PMID 9638695
- [Background] Michaelides PL, Wilson SG. An autogenous gingival graft technique. Int J Periodontics Restorative Dent. 1994 Apr;14(2):112-25. PMID 7928128
- [Background] Okuda K, Kawase T, Momose M, Murata M, Saito Y, Suzuki H, Wolff LF, Yoshie H. Platelet-rich plasma contains high levels of platelet-derived growth factor and transforming growth factor-beta and modulates the proliferation of periodontally related cells in vitro. J Periodontol. 2003 Jun;74(6):849-57. doi: 10.1902/jop.2003.74.6.849. PMID 12886996
- [Background] Paolantonio M, Dolci M, Esposito P, D'Archivio D, Lisanti L, Di Luccio A, Perinetti G. Subpedicle acellular dermal matrix graft and autogenous connective tissue graft in the treatment of gingival recessions: a comparative 1-year clinical study. J Periodontol. 2002 Nov;73(11):1299-307. doi: 10.1902/jop.2002.73.11.1299. PMID 12479634
- [Background] Petrungaro P. Platelet-rich plasma for dental implants and soft-tissue grafting. Interview by Arun K. Garg. Dent Implantol Update. 2001 Jun;12(6):41-6. No abstract available. PMID 11993379
- [Background] Pini-Prato G, Baldi C, Pagliaro U, Nieri M, Saletta D, Rotundo R, Cortellini P. Coronally advanced flap procedure for root coverage. Treatment of root surface: root planning versus polishing. J Periodontol. 1999 Sep;70(9):1064-76. doi: 10.1902/jop.1999.70.9.1064. PMID 10505810
- [Background] Roccuzzo M, Bunino M, Needleman I, Sanz M. Periodontal plastic surgery for treatment of localized gingival recessions: a systematic review. J Clin Periodontol. 2002;29 Suppl 3:178-94; discussion 195-6. doi: 10.1034/j.1600-051x.29.s3.11.x. PMID 12787218
- [Background] Tozum TF, Demiralp B. Platelet-rich plasma: a promising innovation in dentistry. J Can Dent Assoc. 2003 Nov;69(10):664. PMID 14611717
- [Background] Wennstrom JL, Zucchelli G. Increased gingival dimensions. A significant factor for successful outcome of root coverage procedures? A 2-year prospective clinical study. J Clin Periodontol. 1996 Aug;23(8):770-7. doi: 10.1111/j.1600-051x.1996.tb00608.x. PMID 8877664
- [Background] Zucchelli G, Clauser C, De Sanctis M, Calandriello M. Mucogingival versus guided tissue regeneration procedures in the treatment of deep recession type defects. J Periodontol. 1998 Feb;69(2):138-45. doi: 10.1902/jop.1998.69.2.138. PMID 9526912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were selected from the outpatient clinic,Faculty of Dentistry, Cairo University between 30/09/2017 and 1/08/ 2019 Patients >18 Periodontally and systemically healthy Miller class I or II buccal recession defects Presence of identifiable CEJ Clinical indication and/or patient request for recession coverage.
Pre-assignment Details: 5 patients were excluded for not meeting inclusion criteria
Groups:
- CAF+SCTG+PRF: Intervention: surgical procedure consisting of coronally advanced flap + SCTG +PRF membrane
  Patients with class I or II gingival recession will receive treatment that consists of coronally advanced flap (CAF) with subepithelial connective tissue graft (SCTG) and platelet rich fibrin membrane(PRF)
- CAF+SCTG: Patients with class I or II gingival recession will receive treatment that consists of CAF+SCTG (control group)
  CAF +SCTG: the use of coronally advanced flap (CAF) with sub-epithelial connective tissue graft (SCTG) from the palate to cover gingival recession
Period: Overall Study
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
Started | 14 | 14
Completed | 14 (6 months follow-up) | 14 (6 months follow-up)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CAF+SCTG+PRF: Intervention group : surgical procedure consisting of coronally advanced flap + SCTG +PRF membrane
  Patients with class I or II gingival recession will receive treatment that consists of coronally advanced flap (CAF) with subepithelial connective tissue graft (SCTG) and platelet rich fibrin membrane(PRF)
- Total: Total of all reporting groups
Arm/Group | CAF+SCTG+PRF | CAF+SCTG | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white non hispanic | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  Egypt | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Recession Depth
Description: measured from the cemento-enamel junction to the margin of the gingiva at the mid-buccal point of the teeth at basline, 3 months and 6 months. It is recorded in millimeters (mm) with lower values mean better outcome.
Time Frame: baseline-3 months-6 months
Measure: Median (Full Range); unit: length in millimeters
Groups:
- Intervention: CAF+SCTG+PRF: Intervention group : surgical procedure consisting of coronally advanced flap + SCTG +PRF membrane
  Patients with class I or II gingival recession will receive treatment that consists of coronally advanced flap (CAF) with subepithelial connective tissue graft (SCTG) and platelet rich fibrin membrane(PRF)
- Control Group:CAF+SCTG: Patients with class I or II gingival recession will receive treatment that consists of CAF+SCTG (control group)
  CAF +SCTG: the use of coronally advanced flap (CAF) with sub-epithelial connective tissue graft (SCTG) from the palate to cover gingival recession
Arm/Group | Intervention: CAF+SCTG+PRF | Control Group:CAF+SCTG
Number analyzed (Participants) | 14 | 14
length in millimeters
  baseline | 2 [1 to 4] | 2 [2 to 4]
  3 months | 0 [0 to 1] | 0 [0 to 1]
  6 months | 0 [0 to 1] | 0 [0 to 1]

2. Secondary Outcome: Recession Width
Description: It was measured as the distance from mesial and distal papillae along the CEJ. It is recorded in millimeters (mm) where lower values means a better outcome.
Time Frame: baseline-3 months-6 months
Measure: Median (Full Range); unit: length in millimeters (mm)
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
Number analyzed (Participants) | 14 | 14
length in millimeters (mm)
  baseline | 1.5 [1 to 3] | 2 [1 to 3]
  3 months | 0 [0 to 1] | 0 [0 to 1]
  6 months | 0 [0 to 1] | 0 [0 to 1]

3. Secondary Outcome: Root Coverage Gain
Description: (preoperative vertical recession - postoperative vertical recession/preoperative vertical recession) x 100.
Time Frame: at 6 months
Measure: Mean (Standard Deviation); unit: percentage of root coverage
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
Number analyzed (Participants) | 14 | 14
percentage of root coverage | 92.9 (18.2) | 91.6 (17.1)

4. Secondary Outcome: Probing Depth
Description: measured from the gingival margin to the base of the pocket probe at the midbuccal point of the teeth. Its is recorded in millimeters (mm) where lower values mean better outcome.
Time Frame: baseline-3 months-6 months
Measure: Mean (Standard Deviation); unit: length in millimeters(mm)
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
Number analyzed (Participants) | 14 | 14
length in millimeters(mm)
  baseline | 1.71 (0.47) | 1.5 (0.65)
  3 months | 1.07 (0.27) | 1.07 (0.27)
  6 months | 1.07 (0.27) | 1.21 (0.27)

5. Secondary Outcome: Clinical Attachment Level
Description: measured from the CEJ to the base of the sulcus at the midbuccal point of the teeth. Its is recorded in millimeters (mm).
Time Frame: baseline-3 months-6 months
Measure: Mean (Standard Deviation); unit: length in millimeters(mm)
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
Number analyzed (Participants) | 14 | 14
length in millimeters(mm)
  baseline | 3.79 (0.97) | 4 (0.78)
  3 months | 2.14 (0.66) | 2.29 (0.73)
  6 months | 2 (0.69) | 2.07 (0.62)

6. Secondary Outcome: Gingival Biotype
Description: under local anesthesia from 3 mm below the gingival margin trans-gingivally piercing tissues horizontally, perpendicular to the long axis of the tooth until it contacts bone. Its is recorded in millimeters (mm) where higher values mean better outcome.
Time Frame: baseline-3 months-6 months
Measure: Median (Full Range); unit: length in millimeters(mm)
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
Number analyzed (Participants) | 14 | 14
length in millimeters(mm)
  baseline | 1 [1 to 1] | 1 [1 to 1]
  3 months | 3 [2 to 3] | 2.5 [2 to 3]
  6 months | 3 [2 to 4] | 3 [2 to 4]

7. Secondary Outcome: Width of Keratinized Gingiva
Description: from the margin of the gingiva to the mucogingival junction at the midbuccal point of the teeth. Its is reported in millimeters where higher values mean better outcome.
Time Frame: baseline-3 months-6 months
Measure: Mean (Standard Deviation); unit: length in millimeters(mm)
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
Number analyzed (Participants) | 14 | 14
length in millimeters(mm)
  baseline | 2.36 (0.63) | 2.64 (0.74)
  3 months | 3.64 (1.08) | 3.71 (0.73)
  6 months | 3.86 (1.03) | 4.14 (0.86)

8. Secondary Outcome: Patient Satisfaction
Description: printed yes/ no questionnaire with 3 questions:
  1. would you do this surgery again?
  2. would you recommend this treatment to others?
  3. are you satisfied with the results?
Time Frame: questionnaire given to the patient 6 months after the surgery
Measure: Number; unit: percentage of patients satisfied
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
Number analyzed (Participants) | 14 | 14
percentage of patients satisfied | 71.4 | 64.3

9. Secondary Outcome: Root Coverage Esthetic Score (RES)
Description: The RES system evaluates 5 variables 6 months after surgery: Zero, 3, or 6 points are used for the evaluation of the position of the gingival margin (GM). A score of 0 or 1 point is used for each of the following variables: marginal tissue contour (MTC), soft tissue texture (STT), mucogingival junction (MGJ) alignment, and gingival color (GC). the points are then summed up to obtain one figure representing the RES.
  minimum value:0 maximum value: 10 which means better outcome for RES
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
Number analyzed (Participants) | 14 | 14
score on a scale | 9.43 (1.09) | 9.29 (1.27)

10. Secondary Outcome: Post Operative Pain
Description: Numerical Rating Scale (NRS) with numbers from 0 to 10 ('no pain' to 'worstpain imaginable') for the first 2 weeks postoperatively
Time Frame: after 2 weeks from surgery
Measure: Median (Full Range); unit: score on a scale
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
Number analyzed (Participants) | 14 | 14
score on a scale | 9 [7 to 10] | 8.5 [5 to 10]

ADVERSE EVENTS:
Time Frame: 6 months from the surgical procedure
Description: mortality, severe bleeding
Arm/Group | CAF+SCTG+PRF | CAF+SCTG
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT03199118/Prot_SAP_000.pdf